CLINICAL TRIAL: NCT07377240
Title: Study of Obstacles and Barriers to Changing Risky Eating Behaviors in Families of Children With Severe Early Childhood Caries (SECC): a Qualitative Approach (QUALIKIDS)
Brief Title: Study of Obstacles and Barriers to Changing Risky Eating Behaviors in Families of Children With Severe Early Childhood Caries (QUALIKIDS).
Acronym: QUALIKIDS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RNI 2025 COLLADO; 2025-A02056-43 (Other: ANSM)
Record Dates: First submitted 2026-01-13; First posted 2026-01-29 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Early Childhood Caries
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interview (Other)
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — Semi-structured, face-to-face interviews

SUMMARY:
Dental caries is the most common chronic disease in children, and its early form-Early Childhood Caries (ECC)-which particularly affects children under the age of six, represents a major public health problem worldwide. This disease has a negative impact on the quality of life of affected children and their families, and leads to significant functional and developmental consequences. Moreover, due to their young age, these children require specialized care and adapted treatment procedures, particularly the use of general anesthesia (GA) for comprehensive oral rehabilitation.

This conservative therapeutic approach improves the quality of life and orofacial functions of the children concerned, particularly their masticatory ability. However, there remains a significant rate of caries recurrence within the year following treatment. This is largely due to the difficulty families face in changing the dietary habits that contribute to the disease, such as the frequent consumption of sugar-rich foods in all their forms. These families are often bio-psycho-socially vulnerable and have a low level of oral health literacy. They also tend to show lower adherence to preventive measures (oral hygiene practices and regular dental check-ups for children) as well as to the health education and therapeutic interventions proposed to them.

In order to stabilize dental caries in these children, prevent repeated procedures due to recurrent caries, and offer interventions tailored to their needs, it is essential to better understand why oral health behaviors are so difficult to change within these families. This study aims to adopt a qualitative approach to explore the obstacles and barriers to modifying etiological behaviors, particularly dietary behaviors, in families of young children with severe ECC treated under general anesthesia in the specialized care unit of Handiconsult ARA Ouest (CHU Estaing Clermont-Ferrand - CH Riom). Semi-structured, face-to-face interviews conducted with one or both parents will investigate the different dimensions of this issue. A subgroup analysis will compare the factors influencing the adoption of oral health-promoting habits in families of children with and without associated developmental disorders.

DETAILED DESCRIPTION:
The recruitment of participating parents is carried out by one of the dental practitioners who sees families during preoperative consultations (specialized dental care unit of the Handiconsult ARA Ouest program, Estaing Clermont-Ferrand University Hospital, or Riom Hospital).

The investigator who welcomes the family on the first day invites the parents to participate in the study, provides oral and written information on the nature and conduct of the study, and answers any questions they may have. If the parent(s) express an interest in participating in the study, their non-opposition is recorded.

To help encourage open discussion, another investigator conducts the recorded interviews as described above. After seeing the parent off, the investigator also writes an interview report summarizing the general course and circumstances of the interview, a summary of the information obtained for each topic, the key points from the interview, the elements to be repeated or modified for the next interview with another parent, and the exchanges or information gathered after the end of the interview.

A verbatim transcript is produced by hand after the interview, while listening to the recording, ensuring that all identifying information (e.g., names, places, identity of the healthcare team) is removed. Only the interview number (in order) is noted on the verbatim transcript. These audio recordings are destroyed within 15 days of transcription.

Subsequently, as the transcriptions are completed, a thematic analysis by coding is carried out by two independent investigators with the assistance of the CROC scientific collaborator. The transcripts will first be read by each investigator. Qualitative data analysis will then be performed using a thematic framework derived from the literature and developed during the analysis process. Continuous data analysis will be used, and the study will be considered complete when saturation is reached, i.e., when no new concepts are recorded.

ELIGIBILITY:
Inclusion Criteria:

* All parents of children under 6 years of age with CPE-S, consulting the specialized dental care unit as part of the Handiconsult ARA Ouest program for complete conservative oral rehabilitation under general anesthesia
* Verbal agreement from the participant to take part in the study and for audio recording
* Parents who understand and speak French.

Exclusion Criteria:

* Parents of children in foster care.
* Parents under judicial protection, guardianship, or conservatorship.
* Parents who refuse to participate in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Nature and relative frequency of barriers to changing dietary behaviors that cause early childhood caries | day 1
  Identification after analysis of comments collected during a semi-structured interview with one or both parents, for the various topics covered in the interview guide.

SECONDARY OUTCOMES:
Changes in the family's daily life related to managing early tooth decay | day 1
The difficulties encountered by families in accessing appropriate oral health care | day 1
Parents' perceptions of the appropriateness of general anesthesia for their child's dental care and the associated risks | day 1
The type, frequency, and context of the child's consumption of sugary foods, particularly between meals. | day 1
Changes in eating habits implemented since the diagnosis of CPE and difficulties encountered | day 1
The frequency and quality of tooth brushing and other preventive measures in place since the diagnosis of CPE | day 1
Parents' intrinsic or extrinsic motivations for changing habits | day 1
Families' expectations regarding the role of healthcare professionals in managing the disease | day 1
Requests expressed in terms of resources or support | day 1
The nature of the support measures that could be appropriate to parents' requests. | day 1

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Collado, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France